CLINICAL TRIAL: NCT06443671
Title: Neoadjuvant Fruquintinib Plus Tislelizumab Combined With mCapeOX Versus CapeOX for Mid-high pMMR/MSS Locally Advanced Rectal Cancer: A Prospective, Open-label, Multicenter, Randomized Controlled Trial
Brief Title: Neoadjuvant Fruquintinib Plus Tislelizumab Combined With mCapeOX Versus CapeOX for Mid-high pMMR/MSS Locally Advanced Rectal Cancer
Acronym: PKUCH-R09
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH-R09
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer
Keywords: local advanced rectal cancer; neoadjuvant chemotherapy; pMMR/MSS; Furoquinib and Tislelizumab; CapeOX
MeSH Terms: conditions — Rectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CapeOX group (Active Comparator): Receiving CapeOX treatment for up to four cycles before surgery:
  Capecitabine: 1000mg/m2, BID, PO, D1-14, Q3W; Oxaliplatin: 130 mg/m2, intravenous drip for 0-2 hours, D1, Q3W.
  Interventions: Drug: CapeOX
- Fruquintinib and Tislelizumab combined with mCapeOX (Experimental): Receiving Fruquintinib plus Tislelizumab combined with mCapeOX treatment for up to four cycles before surgery:
  Fruquintinib: 3mg/d, QD, PO, Use for 2 weeks, stop for 1 week, Q3W; Tislelizumab: 200mg, D1, Intravenous infusion, Q3W; Capecitabine: 825mg/m2, BID, PO, D1-14, Q3W; Oxaliplatin: 100 mg/m2, intravenous drip for 0-2 hours, D1, Q3W.
  Interventions: Drug: Fruquintinib and Tislelizumab combined with mCapeOX

INTERVENTIONS:
Drug: CapeOX — Receiving CapeOX treatment for up to four cycles before surgery:
  Capecitabine: 1000mg/m2, BID, PO, D1-14, Q3W; Oxaliplatin: 130 mg/m2, intravenous drip for 0-2 hours, D1, Q3W.
  Arms: CapeOX group
Drug: Fruquintinib and Tislelizumab combined with mCapeOX — Receiving Fruquintinib plus Tislelizumab combined with mCapeOX treatment for up to four cycles before surgery:
  Fruquintinib: 3mg/d, QD, PO, Use for 2 weeks, stop for 1 week, Q3W; Tislelizumab: 200mg, D1, Intravenous infusion, Q3W; Capecitabine: 825mg/m2, BID, PO, D1-14, Q3W; Oxaliplatin: 100 mg/m2, intravenous drip for 0-2 hours, D1, Q3W.
  Arms: Fruquintinib and Tislelizumab combined with mCapeOX

SUMMARY:
The goal of this clinical trial is to learn if neoadjuvant Fruquintinib and Tislelizumab combined with mCapeOX works to treat mid-high pMMR/MSS locally advanced rectal cancer patients compared with CapeOX. It will also learn about the safety of neoadjuvant Fruquintinib and Tislelizumab combined with mCapeOX. The main questions it aims to answer are:

* Does neoadjuvant Fruquintinib and Tislelizumab combined with mCapeOX improve the pCR rate of mid-high pMMR/MSS locally advanced rectal cancer patients?
* What medical problems do participants have when receiving neoadjuvant Fruquintinib and Tislelizumab combined with mCapeOX? Researchers will compare Fruquintinib and Tislelizumab combined with mCapeOX to CapeOX to see if neoadjuvant Fruquintinib and Tislelizumab combined with mCapeOX works to treat mid-high pMMR/MSS locally advanced rectal cancer patients.

Participants will:

* Receive Fruquintinib and Tislelizumab combined with mCapeOX or CapeOX before surgery up to 4 cycles
* Receive radical operations and three years follow-up
* Keep a diary of their postoperative pathology results and survival

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study and signed an informed consent form;
* Age: 18-75 years old (including 18 and 75 years old), regardless of gender;
* Histologically confirmed rectal adenocarcinoma; Immunohistochemistry suggests pMMR, or PCR suggests MSS type patients;
* The tumor location meets the following criteria:

  1. Colonoscopy or digital examination shows that the distance from the lower edge of the tumor to the anus is 6-15cm or more than 4cm from the ARJ;
  2. MRI/CT determines that the lower edge of the tumor or the lower edge of the invading part is not higher than the sacral promontory pubic line;
* Preoperative staging meets the following conditions:

  1. Preoperative staging of tumor infiltration breaking through the intestinal muscle layer (T3) or above or accompanied by periintestinal lymph node metastasis;
  2. Non invasion of the intrinsic fascia of the rectum (MRF -);
  3. No swelling observed in lateral lymph nodes (short diameter not exceeding 7mm)
  4. There is no clear evidence of distant metastasis, and R0 resection is expected to be feasible after treatment; *Baseline partial phase method: Rectal T2/DWI MR or Abdominal Pelvic CT or PET/CT or PET/MRI;
* Have not received any anti-tumor treatment for rectal cancer in the past, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc;
* ECOG score: 0-1 points;
* Able to swallow tablets and capsules normally;
* The plan is to complete the entire process of neoadjuvant therapy and undergo surgical resection;
* The main organs and bone marrow function are basically normal (no blood components or cell growth factors were used within 14 days before enrollment):

  1. Blood routine: Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 90g/L;
  2. International standardized ratio (INR) ≤ 1.5 x Upper limit of normal value (ULN), and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
  3. Liver function: Total bilirubin ≤ 1.5 x ULN, ALT/AST ≤ 2.5 x ULN；
  4. Renal function: serum creatinine ≤ 1.5 x ULN, and creatinine clearance rate (CCr) ≥ 50mL/min;
* Women of childbearing age must undergo a serum pregnancy test within 14 days before treatment, and the result is negative; Qualified patients with fertility (male and female) must agree to use reliable contraceptive methods (hormone or barrier methods or abstinence, etc.) with their partners during the trial period and at least 6 months after the last medication.

Exclusion Criteria:

* Have a history of allergies to any anti-angiogenic targeted drugs, any components of monoclonal antibodies, capecitabine, oxaliplatin, or other platinum-based drugs in the past;
* Preoperative evidence suggests distant metastasis (including lymph node metastasis in the iliac foramen area) Metastasis of aortic lymph nodes and retroperitoneal lymph nodes above the root level of IMA; In addition to clear liver lung metastasis, liver lung nodules with unknown properties should also be excluded;
* Symptoms of incomplete or complete intestinal obstruction; Or preoperative colonoscopy may indicate narrowing of the intestinal lumen circumference; Or if the tumor is too large, colonoscopy cannot pass through the tumor;
* Those who are currently using immunosuppressive agents, systemic or absorbable local hormone therapy to achieve immunosuppressive effects (dosage>10mg/day prednisone or other therapeutic hormones), and continue to use them within 2 weeks prior to enrollment;
* Receive attenuated live vaccines within 4 weeks prior to the first use of the study drug;
* Any active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or complete remission of childhood asthma in adulthood without any intervention can be included; subjects with asthma requiring medical intervention with bronchodilators cannot be included);
* Other malignant tumors in the past 5 years (excluding skin basal cell or squamous cell carcinoma, cervical carcinoma in situ, breast cancer, thyroid papillary carcinoma and small kidney carcinoma that are clinically cured after proper treatment (OS>5 years));
* Congenital or acquired immune deficiency (such as HIV infected persons), or active hepatitis (hepatitis B: HBsAg positive and HBV DNA ≥ 104 copies/ml; hepatitis C: HCV antibody positive and HCV RNA>1 × 103 copies/ml);
* Have uncontrolled clinical symptoms or diseases of the heart, such as: (1) NYHA grade 2 or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention;
* Suffering from hypertension and unable to achieve good control through antihypertensive drug treatment (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
* Active or uncontrolled severe infections (≥ CTCAE level 2 infection);
* Urinary routine indicates that urine protein is ≥ 2+, and the 24-hour urine protein content is>1.0g;
* Known genetic or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation dysfunction, thrombocytopenia, splenic hyperfunction, etc.) or undergoing thrombolytic or anticoagulant therapy;
* The patient currently has digestive tract diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectable tumors, or other conditions determined by the researcher that may cause gastrointestinal bleeding or perforation;
* Patients with significant evidence of bleeding tendency or medical history within the 3 months prior to enrollment (bleeding>30 mL within 3 months, vomiting blood, black stool, and rectal bleeding), hemoptysis (fresh blood>5 mL within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months;
* Pregnant (positive pregnancy test before medication) or breastfeeding women;
* According to the judgment of the researchers, the subjects may have other situations that may affect the results of the study or cause the study to be forced to stop midway, such as drug abuse, serious illnesses (including mental illnesses such as seizures), and other medical, psychological, or social conditions that may endanger patient safety and compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response(pCR) rates | 10 days after surgery
  Pathological complete response(pCR) rates are defined as no viable tumor cells remaining in the primary tumor and lymph nodes (ypT0N0), that is, subjects with level 0 of the AJCC 8th edition Tumor Regression Grading (TRG) scoring system proportion.

SECONDARY OUTCOMES:
Adverse events (AEs) | From the beginning to the 21st day after the end of neoadjuvant treatment
  Adverse events (AEs) refer to adverse medical events that occur after clinical trial subjects receive a drug, but are not necessarily causally related to the treatment. AE can be any adverse and unexpected symptoms, signs, laboratory test abnormalities or diseases, etc., including at least the following situations: 1) Pre-existing medical conditions/diseases (before entering clinical trials) will be recorded as adverse events only if they worsen after starting to use the trial drug (including worsening of symptoms, signs, and laboratory test abnormalities); 2) Any new AE: any new adverse medical condition (including symptoms, signs, newly diagnosed diseases); 3) Abnormal clinically significant laboratory test results. Diagnostic or therapeutic invasive (such as surgery) and non-invasive procedures should not be reported as AEs, but when the disease condition that causes the procedures meets the definition of AE, they should be reported.
Major Pathologic Response(MPR) | 10 days after surgery
  MPR: The proportion of residual viable tumor cells in the postoperative specimen in the tumor bed is less than or equal to 10%.
3-year event-free survival (EFS) rate | 36 months after randomization
  EFS is defined as the time from randomization to the occurrence of any of the following events, whichever occurs first: tumor disease progression on imaging as assessed by RECIST 1.1; tumor recurrence, including local recurrence or distant recurrence, as assessed on imaging or tissue biopsy transfer; death from any cause.
3-year overall survival (OS) rate | 36 months after randomization
  OS is defined as the time between the date of randomization and death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No